CLINICAL TRIAL: NCT07022600
Title: Erector Spinae Plane Block and Its Impact on Postoperative Diaphragmatic Dysfunction in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy, A Double-blind Randomized Control Trial.
Brief Title: Erector Spinae Plane Block and Its Impact on Postoperative Diaphragmatic Dysfunction in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical acre, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ESPB and its impact on DD
Record Dates: First submitted 2025-05-12; First posted 2025-06-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Diaphragmatic Dysfunction
Keywords: erector spinae block; diaphragmatic dysfunction; morbidly obese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae group (Active Comparator): Patients will receive erector spinae block
  Interventions: Device: Diaphragmatic ultrasound
- Control group (Placebo Comparator): Patients will receive bilateral sham ultrasound-guided ESPB
  Interventions: Device: Diaphragmatic ultrasound

INTERVENTIONS:
Device: Diaphragmatic ultrasound — diaphragmatic excursion will be conducted at baseline and at 2 and 24 hours postoperatively

SUMMARY:
postoperative diaphragmatic dysfunction is critical especially in morbidly obese patients

DETAILED DESCRIPTION:
Investigators aimed to evaluate the impact of erector spinae plane block on the incidence of postoperative diaphragmatic dysfunction in morbidly obese patients (Body mass index more than or equal 40)

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese (body mass index> 40)
* undergoing sleeve gastrectomy

Exclusion Criteria:

* allergy to bupivacaine
* respiratory comorbidities
* preoperative diaphragmatic dysfunction
* Patient refusal
* inability to adequately visualize diaphragm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of diaphragmatic dysfunction in both groups | baseline and 2 hours after surgery
  postoperative diaphragmatic excursion 10 mm at 2 hours after surgery

SECONDARY OUTCOMES:
Forced expiratory volume at one second | at baseline, 2 and 24 hours postoperatively
  FEV1 (in liter)
numeric rating scale | at 24 hours after surgery
  score from zero to 10
Forced vital capacity (in Liter) | at baseline, 2 hours, and 24 hours after surgery
  FVC (in liter)
Peak expiratory flow rate (Liter/sec) | baseline, 2 hours, and 24 hours
  PEFR (Liter/sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to privacy concerns, regulatory restrictions, and informed consent limitations.

REFERENCES:
- [Background] Helmy MA, Hasanin A, Milad LM, Mostafa M, Hamimy WI, Muhareb RS, Raafat H. Ability of parasternal intercostal muscle thickening fraction to predict reintubation in surgical patients with sepsis. BMC Anesthesiol. 2024 Aug 22;24(1):294. doi: 10.1186/s12871-024-02666-8. PMID 39174907
- [Background] Yildiz M, Kozanhan B, Iyisoy MS, Canitez A, Aksoy N, Eryigit A. The effect of erector spinae plane block on postoperative analgesia and respiratory function in patients undergoing laparoscopic cholecystectomy: A double-blind randomized controlled trial. J Clin Anesth. 2021 Nov;74:110403. doi: 10.1016/j.jclinane.2021.110403. Epub 2021 Jul 26. PMID 34325186
- [Background] Helmy MA, Magdy Milad L, Osman SH, Ali MA, Hasanin A. Diaphragmatic excursion: A possible key player for predicting successful weaning in patients with severe COVID-19. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100875. doi: 10.1016/j.accpm.2021.100875. Epub 2021 Apr 30. No abstract available. PMID 33940248
- [Background] Helmy MA, Mostafa L, El-Zayyat NS, Ali MA, Sabry R. Impaired diaphragmatic excursion following magnesium sulfate administration in patients with preeclampsia with severe features: a prospective observational study. Int J Obstet Anesth. 2025 May;62:104347. doi: 10.1016/j.ijoa.2025.104347. Epub 2025 Feb 28. PMID 40101564
- [Background] Mostafa SF, Abdelghany MS, Abu Elyazed MM. Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Laparoscopic Bariatric Surgery: A Prospective Randomized Controlled Trial. Pain Pract. 2021 Apr;21(4):445-453. doi: 10.1111/papr.12975. Epub 2021 Jan 22. PMID 33295128